CLINICAL TRIAL: NCT04034082
Title: Effect of Intermittent Hypoxia Therapy on Functional Capacity in Geriatric Cardiac Patients With Functional Impairment During a Cardiac Rehabilitation Program: a Pilot Study
Brief Title: Intermittent Hypoxia Therapy in Cardiac Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2233CE
Record Dates: First submitted 2019-07-22; First posted 2019-07-26 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2019-07

CONDITIONS: Cardiovascular Disease; Exercise; Hypoxia
Keywords: cardiovascular disease; rehabilitation; exercise
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IHT group (Experimental): Intermittent hypoxia therapy on top of the conventional phase 2 in-hospital rehabilitation program
  Interventions: Device: Intermittent hypoxia therapy; Other: Conventional phase 2 cardiac rehabilitation programme
- Conventional group (Active Comparator): Conventional phase 2 in-hospital rehabilitation program
  Interventions: Other: Conventional phase 2 cardiac rehabilitation programme

INTERVENTIONS:
Device: Intermittent hypoxia therapy — Intermittent Hypoxic Therapy (further referred to as IHT). A typical IHT session consists of repeated short-term moderate hypoxia (down to 10 vol.% O2), interrupted by brief periods of reoxygenation. These periods of recovery could be either normoxic (21 vol.% O2, Hypoxia-Normoxia mode) or hyperoxic (30-35 vol.% O2, Hypoxia-Hyperoxia mode, further referred to as IHHT). The gas mixtures are supplied to a patient via facial mask.
  Arms: IHT group
Other: Conventional phase 2 cardiac rehabilitation programme — The core components of a Phase 2 in-hospital cardiac rehabilitation program include: 1) patient assessment with medical control to promote clinical stabilization and optimization of pharmacologic treatment; 2) physical activity counselling; 3) prescription of an individualized exercise training; 4) diet/nutritional counselling; 5) weight control management; 6) Lipid management; 7) blood pressure monitoring and management; 8) smoking cessation; 9) vocational support; 10) psychosocial management..

SUMMARY:
This is a randomized control pilot study to assess the effect of intermittent hypoxia therapy on functional capacity vs conventional care in old patients with functional impairment admitted to a Phase 2 in-hospital cardiac rehabilitation program.

DETAILED DESCRIPTION:
Because the improvement of exercise tolerance reduces mortality in elderly patients affected by cardiovascular disease, intermittent hypoxia therapy (IHT) - defined as repeated episodes of hypoxia interspersed with normoxic periods delivered by an ad hoc device - might be a valuable tool to be associated to structured cardiac rehabilitation (CR) interventions.

The present study is a pilot, monocentric, randomized (randomization ratio 1:1), parallel group study to assess the effect of IHT on functional capacity vs conventional care in old patients with functional impairment admitted to a phase 2 in-hospital cardiac rehabilitation program.

The study will enroll cardiac patients of both genders, ≥ 75 years and with a functional impairment assessed by a Short Physical Performance Battery (SPPB) score < 7.

The effect of IHT on functional capacity will be evaluated on top of the conventional multidisciplinary CR intervention, by means of SPPB score variation; variations in quality of life and cognitive status will also be evaluated as secondary goals of the study.

The total amount of IHT sessions per patient will be 10, 1 per day over 2 weeks, the duration of each single procedure will be 45 min and the Hypoxic O2 conc.% will be 14-10. The study was approved by local ethic committee.

ELIGIBILITY:
Inclusion Criteria:

* Admission to a Phase 2 in-hospital cardiac rehabilitation program because of a recent index event;
* Provision of signed and dated informed consent form;
* Age ≥ 75 years;
* Basic venous blood oxygen saturation (SpO2) level > 93% measured at the fingertip;
* SPPB score < 7;
* New York Heart Association (NYHA) Class I-III.

Exclusion Criteria:

* Inability to give informed consent (diminished understanding or comprehension);
* Age < 75 years;
* SPPB Score ≥ 7;
* NYHA Class IV and/or concomitant i.v. therapy with cardiovascular active drugs;
* Uncontrolled angina pectoris;
* Uncontrolled arterial hypertension;
* Uncontrolled atrial or ventricular arrhythmias;
* Active pericarditis or myocarditis;
* Need of continuous or intermittent O2 therapy;
* Hb < 10 g/dl;
* Severe concomitant non-cardiac diseases such as cancer or any other systemic disease limiting to participate in the study
* Acute inflammatory diseases;
* Acute non-cardiac somatic diseases, or somatic diseases with symptoms of decompensation;
* Currently implanted left ventricular assist device;
* Inability to accept the procedure of breathing via facial mask.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Changes in SPPB score | 30 days
  The Short Physical Performance Battery (SPPB) is a series of physical performance tests used in older persons to assess lower extremity function and mobility.
  Score total: minimum 0 (lowest performance), maximum 12 (highest performance). Three subscales (minimum 0, maximum 4 points each one): balance test, gait speed test, chair stand test.

SECONDARY OUTCOMES:
Changes in distance at the 6-min walking test | 30 days
  6-min walking test is a test for functional evaluation based on walking distance performed by the patient in the time window at the individual walking speed. Score in meters: minimum zero, maximum indefinite
Changes in peak exercise oxygen uptake (peak VO2) | 30 days
  Peak VO2 represents the maximal individualized oxygen consumption at the peak effort, evaluated by means of cardiopulmonary exercise testing, expressed by means of ml of oxygen per Kg of body weight per minute.
Changes in basal blood pressure | 30 days
  Expressed by means of mmHg. Indicator of haemodynamic status.
Changes in basal heart rate | 30 days
  Expressed by means of number of beats per minute. Indicator of haemodynamic status.
Changes in EuroQoL score | 30 days
  European Quality of Life score (EuroQoL). Score: from 0 (lowest condition) to 10 (best condition).
Changes in geriatric depression scale | 30 days
  30 items with relative categorization (1 present; 0 absent). Minimum 0 points (absence of depression), maximum 30 point (highest grade of depression).
Changes in minimental state evaluation | 30 days
  Tool for evaluation of cognitive status in older patients. Minimum score 0 (absence of cognitive impairment), maximum 30 (highest grade of cognitive impairment)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Pedretti, MD, Study Chair — ICS Maugeri care and Research Institute, Pavia, Italy
Locations (1):
- Istituti Clinici Scientifici Maugeri IRCCS, Pavia, Italy